CLINICAL TRIAL: NCT05116384
Title: A Trial to Evaluate Renal Artery Denervation in Addition to Catheter Ablation to Eliminate Atrial Fibrillation
Brief Title: Renal Denervation + PVI vs PVI Alone for Persistent AF
Acronym: ERADICATE-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jonathan Steinberg, Professor of Medicine (adj), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UR ERADICATE-AF II; R34HL153579 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-11-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Pulmonary vein isolation (Active Comparator): Electrical isolation by cryoballoon of all pulmonary veins
  Interventions: Device: catheter ablation
- Pulmonary vein isolation + renal artery denervation (Experimental): After completion of the standard PVI, radiofrequency ablation of bilateral renal arteries
  Interventions: Device: catheter ablation; Device: renal artery denervation

INTERVENTIONS:
Device: catheter ablation — cryo energy via cryoballoon
Device: renal artery denervation — RF energy delivery to multiple sites within each major renal artery
  Arms: Pulmonary vein isolation + renal artery denervation

SUMMARY:
Pulmonary vein isolation (PVI) is the cornerstone of ablation for atrial fibrillation (AF). Increased cardiac sympathetic stimulation can facilitate AF and reduction can be accomplished by renal artery denervation (RDN). The recently completed randomized trial, ERADICATE-AF, convincingly demonstrated that RDN plus PVI resulted in a reduction in recurrent incident AF for uncontrolled hypertensives.

This is a randomized controlled pilot trial, "To Evaluate Renal Artery Denervation in Addition to Catheter Ablation to Eliminate Atrial Fibrillation" (ERADICATE-AF II) to test if RDN plus PVI enhances long-term efficacy vs PVI for persistent AF patients with controlled or without hypertension using implantable loop recordings.

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) is the cornerstone of ablation strategies for atrial fibrillation (AF) and is the only cardio-centric approach consistently shown to be effective for reducing arrhythmia recurrence and improving symptom status. Catheter ablation is superior to medical therapy and current antiarrhythmic drug options are limited, can have significant adverse effects, and are associated with a high arrhythmia recurrence rate, especially for persistent AF. Catheter ablation is now commonly prescribed for symptomatic AF patients who do not respond to medications and carries a class II indication. Thousands of patients undergo catheter ablation in the US each year. Nonetheless, even with technical advances, PVI has a recognized and significant rate of short- and long-term failure, and often requires multiple procedures to establish success.

The mechanisms of AF are diverse, but increased central sympathetic outflow and efferent cardiac sympathetic nerve stimulation can lead to enhanced automaticity and triggered activity, and thus contribute to the development and perpetuation of AF. Reduction in cardiac sympathetic input has been proposed as a logical adjunctive approach to PVI but its technical application via cardiac ablation (targeting autonomic ganglia) has had mixed results at best.

The therapeutic objective of lesser cardiac sympathetic stimulation can be potentially accomplished by renal artery denervation (RDN), a technique originally developed for the treatment of resistant hypertension. RDN's potential for antiarrhythmic effect may be mediated by reduced central nervous sympathetic output and is exemplified by a decrease in whole-body norepinephrine spillover and muscle-sympathetic nerve activity.

The recently completed large-scale, randomized, multicenter, single-blind clinical trial, ERADICATE-AF, demonstrated that RDN plus PVI resulted in a relative 43% reduction (absolute change, 15%; P < 0.001) in recurrent incident AF during one year of follow-up. The trial enrolled > 300 patients with paroxysmal AF referred for ablation, all with poorly controlled hypertension despite medication. There was no difference in complications between the 2 groups, and the procedure with RDN was only lengthened by about 24 minutes.

The trial results suggested that a strategy of reducing cardiac autonomic input is an effective antiarrhythmic approach, in line with many preclinical models. It also represents a paradigm of the potential for complementary noncardiac ablation that is effective and safe when coupled with PVI. Until now, this approach has only been tested in patients with resistant and/or poorly controlled hypertension.

A randomized controlled pilot clinical trial has been proposed: "A Trial to Evaluate Renal Artery Denervation in Addition to Catheter Ablation to Eliminate Atrial Fibrillation" (ERADICATE-AF II), to test the hypothesis that RDN in addition to PVI enhances long-term antiarrhythmic efficacy in comparison to PVI alone for patients with persistent AF with controlled hypertension or without hypertension in a multicenter, single-blinded, longitudinal randomized clinical trial. The trial will be advantaged by performing implantable loop recordings (ILR) in all patients, which will facilitate the calculation of AF burden, now recognized as a powerful predictor of clinical outcome. With successful completion of this pilot program, we hope to launch a large-scale trial with cardiovascular and death events as endpoints.

The primary aim of the study:

To determine if patients with persistent AF with controlled hypertension or without hypertension who are referred for catheter ablation (PVI) and undergo adjunctive RDN have reduced AF burden at 12 months in comparison to patients who undergo only PVI

The following secondary aims will be tested:

In patients with persistent AF with controlled hypertension or without hypertension who are referred for catheter ablation (PVI) and undergo adjunctive RDN relative to patients who undergo only PVI:

1. To assess safety, blood pressure and autonomic nervous system outcomes

   1. Procedural complications rates
   2. Postural blood pressure changes over time
   3. Ambulatory blood pressure monitor results
   4. Cardiac sympathetic nervous system modulation
2. To evaluate clinical end points

   1. Frequency of progression to recurrent persistent AF
   2. Referral for repeat catheter ablation of AF
   3. Need for cardiovascular emergency room visits and hospitalizations
3. To measure effects on quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Symptomatic persistent AF eligible for referral for PVI based on current guidelines1 (persistent AF defined as continuation > 7 days and up to 1 year)
3. No prior history of HTN or HTN controlled on medical therapy (defined as SBP <140 mm Hg and DBP <85 mm Hg)
4. Renal vasculature accessible as determined by pre-procedural renal magnetic resonance angiogram
5. Willingness to undergo ILR placement
6. Willingness to comply with post-procedural follow-up requirements and to sign informed consent.

Exclusion Criteria:

1. Inability to undergo AF catheter ablation (e.g., presence of a left atrial thrombus, contraindication to all anticoagulation)
2. Prior left atrial ablation for an atrial arrhythmia
3. NYHA class IV congestive heart failure or LVEF < 25%
4. Paroxysmal AF, or longstanding persistent AF (duration > 1 year)
5. Coronary revascularization or valve surgery within 3 months
6. Prior valve surgery using a mechanical prosthesis
7. Renal artery anatomy that is ineligible for treatment including:

   1. Predicted inability to access renal vasculature
   2. Main renal arteries < 4 mm in diameter or < 20 mm in length.
   3. Hemodynamically or anatomically significant renal artery abnormality or stenosis
   4. A history of prior renal artery intervention including balloon angioplasty or stenting that precludes a possibility of ablation treatment
   5. Multiple main renal arteries to either kidney
8. An estimated glomerular filtration rate (eGFR) < 45mL/min/1.73m2, using the MDRD calculation
9. Life expectancy <1 year for any medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
AF burden | At 1 year
  The calculated total amount of time in AF after 3-month blanking period

SECONDARY OUTCOMES:
Procedural complications, radiation exposure, and duration | 30 days and 12 months
  Adverse events
BP changes over time | At 0, 1, 3, 6 and 12 months
  Orthostatic BP measurements
BP changes over time | 6 months vs baseline
  Ambulatory BP monitoring
Cardiac sympathetic nervous system modulation | At 0, 1, 3, 6 and 12 months
  Heart rate variability
Cardiac sympathetic nervous system modulation | At 0, 1, 3, 6 and 12 months
  ECG-based biomarker: period repolarization dynamics (beat-to-beat variation of T wave vector)
Quality of life in response to ablation | 6 months vs baseline
  Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT); Overall scores ranging from 0-100 (100 best)
Quality of life in response to ablation | 6 months vs baseline
  Short-Form (SF)-12 questionnaire; Overall scores ranging from 0-100 (100 best)
Number of subject with recurrent atrial fibrillation | From date of randomized procedure to 12 months
  Persistent AF; repeat ablation
Number of subjects with CV hospitalization and/or ER visits | From date of randomized procedure to 12 months
  Clinical events
Total mortality rate | From date of randomized procedure to 12 months
  Death events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Short Hills, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steinberg JS, Shabanov V, Ponomarev D, Losik D, Ivanickiy E, Kropotkin E, Polyakov K, Ptaszynski P, Keweloh B, Yao CJ, Pokushalov EA, Romanov AB. Effect of Renal Denervation and Catheter Ablation vs Catheter Ablation Alone on Atrial Fibrillation Recurrence Among Patients With Paroxysmal Atrial Fibrillation and Hypertension: The ERADICATE-AF Randomized Clinical Trial. JAMA. 2020 Jan 21;323(3):248-255. doi: 10.1001/jama.2019.21187. PMID 31961420